CLINICAL TRIAL: NCT07177209
Title: Describing Prescription Patterns in an Ulcerative Colitis Population and Generating an Updated Ulcerative Colitis Treatment Paradigm
Brief Title: Describing Treatment Patterns and Creating an Updated Treatment Flow in an Ulcerative Colitis Population
Acronym: EFFECT-1LAT
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C5041058
Record Dates: First submitted 2025-08-01; First posted 2025-09-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod; ozanimod; GLPG0634; tofacitinib; vedolizumab; guselkumab; Ustekinumab; risankizumab; Adalimumab; Infliximab; golimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A: Patients within the Lothian IBD registry, approximately 4000 patients, of which 3200 are on conventional therapy.
  Interventions: Drug: Non-Interventional Study
- Cohort B: Patients with uncontrolled inflammation defined as two or more episodes of raised CRP or faecal calprotectin recording 6-24 months post UC diagnosis.
  Interventions: Drug: Non-Interventional Study
- Cohort C: Patients with steroid dependent controlled inflammation defined as normal CRP and faecal calprotectin but the requirement of a dose of steroids between 6-24 months.
  Interventions: Drug: Non-Interventional Study
- Cohort D: Patients with controlled inflammation defined as the absence of steroid requirement or normal CRP or faecal calprotectin 6-24 months post UC diagnosis
  Interventions: Drug: Non-Interventional Study

INTERVENTIONS:
Drug: Non-Interventional Study — As provided in real world practice
  Other Names: etrasimod; ozanimod; upadicitinib; filgotinib; tofacitinib; vedolizumab; guselkumab; ustekinumab; risankizumab; adalimumab; infliximab; golimumab

SUMMARY:
Describing Treatment Patterns and Creating an Updated Treatment Flow in an Ulcerative Colitis Population

DETAILED DESCRIPTION:
Exploring the long-term outcomes of uncontrolled inflammation, and how does early switching to advanced treatments affect disease outcomes and inflammation control in patients with poorly controlled ulcerative colitis.

ELIGIBILITY:
Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Patient enrolled in IBD registry from 2009
2. >18 years at time of diagnosis.
3. Diagnosis of Ulcerative Colitis.
4. Patient data entered during the study period.
5. Minimum duration of data post UC diagnosis (Cohort A: 6 months, Cohort B-D 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Lothian IBD registry (LIBDR) was compiled through a capture-recapture methodology, describes the observed prevalence of IBD in Lothian between 2008 and 2018, and has been maintained as a prospective registry since 1 August 2018 and thus the study period is up to 1st August 2025 (2008 - 2025). The study size is expected to be a defined population of approximately 4000 UC patients, with more than 600 having commenced an advanced therapy. The study period will be from 2008 - 2025.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that achieve early control of inflammation on conventional therapeutics within 6-24 months of UC diagnosis. | 6-24 months from UC diagnosis.
  Proportion of patients that achieve early control of inflammation on conventional therapeutics within 6-24 months of UC diagnosis in the Lothian inflammatory bowel disease registry (LIBDR).
Difference in proportion of patients with inadequate control of inflammation (defined as two or more episodes of raised CRP or faecal calprotectin) treated with conventional therapeutics versus treatment escalation 24 months post UC diagnosis. | 24 months
  Explore the differences in long term outcomes for patients with uncontrolled inflammation, treated with prolonged conventional therapeutics versus treatment escalation up to 24 months for patients with inadequate control of inflammation in the Lothian inflammatory bowel disease registry (LIBDR).

SECONDARY OUTCOMES:
Characterise patient demography at the time of diagnosis and associated co-morbidities and extra-intestinal manifestations of interest. | Baseline demography.
  Characterise patient demography at the time of UC diagnosis and associated co-morbidities and extra-intestinal manifestations of interest in the Lothian inflammatory bowel disease registry (LIBDR).
Map treatment use from conventional therapies to advanced therapies from time of UC diagnosis. | Study period is up to 1st August 2025 (2008 - 2025).
  Map treatment use from from conventional therapies to advanced therapies from time of UC diagnosis in the Lothian inflammatory bowel disease registry (LIBDR).
Change from Baseline in Faecal Calprotectin (Fcal). | Study period is up to 1st August 2025 (2008 - 2025).
  Generate Faecal Calprotectin (Fcal) profile and longitudinal inflammatory response models for patients on conventional therapy in the Lothian inflammatory bowel disease registry (LIBDR).
Change from Baseline in C-Reactive Protein (CRP). | Study period is up to 1st August 2025 (2008 - 2025).
  Generate C-Reactive Protein (CRP) profile and longitudinal inflammatory response models for patients on conventional therapy in the Lothian inflammatory bowel disease registry (LIBDR).
Proportion of patients with colectomies from baseline. | Study period is up to 1st August 2025 (2008 - 2025).
  Assess colectomy rates of patients in the Lothian inflammatory bowel disease registry (LIBDR) with a relevant UC diagnosis.
Proportion of patients with hospitalisations from baseline. | Study period is up to 1st August 2025 (2008 - 2025).
  Assess hospitalisation rates in the Lothian inflammatory bowel disease registry (LIBDR) with a relevant UC diagnosis.
Proportion of patients with advanced therapy (AT) requirements with relevant UC diagnosis. | Study period is up to 1st August 2025 (2008 - 2025).
  Assess advanced therapy (AT) requirements in the Lothian inflammatory bowel disease registry (LIBDR).
Correlate duration of uncontrolled inflammation within first 6-24 months of treatment to long term outcomes as provided in real world evidence practice. | Study period is up to 1st August 2025 (2008 - 2025).
  Duration of uncontrolled inflammation in the Lothian inflammatory bowel disease registry (LIBDR).
Describe the effects of conventional treatment to AT's (etrasimod and tofacitinib) by change from baseline in steroid utilisation. | Study period is up to 1st August 2025 (2008 - 2025).
  Effects of conventional treatment to advanced therapies (AT's) in steroid utilisation in the Lothian inflammatory bowel disease registry (LIBDR).
Change from baseline in control of inflammation (CRP or faecal calprotectin) in patients that are moved from conventional treatments to advanced treatments with a UC diagnosis. | From baseline, study period is up to 1st August 2025 (2008 - 2025).
  Describe the effects of changing from conventional treatment to advanced treatments (etrasimod and tofacitinib) in control of inflammation (CRP or faecal calprotectin) in the Lothian inflammatory bowel disease registry (LIBDR).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Walton Oaks, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.